CLINICAL TRIAL: NCT02212444
Title: The Effectiveness of a Dynamic Elastomeric Fabric Orthoses (DEFO) in the Management of Plantar Fasciitis: A Feasibility Study
Brief Title: Comparing the Effects of Two Foot and Ankle Splints for Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 14/P/051; 14/SW/0116 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-08-04; First posted 2014-08-08 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; dynamic elastomeric fabric orthoses (DEFO); feasibility; Physiotherapy; Musculoskeletal
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic elastomeric fabric orthoses (DEFO) (Experimental): The DEFO will be provided after taking the baseline measures and orthoses measurements at the baseline session ~ 3 weeks later. The orthoses will be supplied via post and used for a period of 12 weeks.
  Interventions: Device: Dynamic elastomeric fabric orthoses (DEFO)
- Off-the-self orthotics (Active Comparator): Off-the-shelf-Orthotics: Patients in the usual care group will be referred for off -the-shelf triplanar orthoses as indicated by a biomechanical assessment of foot posture while standing / walking on visit 1. The off the shelf orthotic will be provided after taking the baseline measures and orthoses measurements at the baseline session ~ 3 weeks later. The orthoses will be supplied via post and used for a period of 12 weeks.
  Interventions: Device: Off -the-shelf triplanar orthoses

INTERVENTIONS:
Device: Dynamic elastomeric fabric orthoses (DEFO) — A patient customised dynamic elastomeric fabric orthoses (DEFO)
  Other Names: DEFO
  Arms: Dynamic elastomeric fabric orthoses (DEFO)
Device: Off -the-shelf triplanar orthoses
  Arms: Off-the-self orthotics

SUMMARY:
Plantar fasciitis (severe pain in the heel) is a common problem that has a significant impact on quality of life. There is some evidence to support the use of orthoses and stretches in the conservative management of plantar fasciitis but current orthotic management may not be optimal. More prolonged stretching with night splints may achieve better results but such splints are clinically not well tolerated. Therefore, there is a potential need to apply prolonged stretching during the day and during dynamic tasks such as walking. This has led to the development of other rigid and semi-rigid splints that have shown promising results in small scale clinical trials. There are disadvantages however with the more rigid bracing and orthoses seen in these types of splints. For example, they are often difficult to accommodate with a person's available shoes; this can be particularly difficult for women and thus limits their compliance with the intervention. Further, more rigid bracing can be uncomfortable during fast walking and running and so limits participation in such activities.

Recently a novel orthotic, a customised dynamic elastomeric fabric orthoses (DEFO), has been developed. Being made from lycra® based materials the sock-like splint is lightweight and discrete, allowing it to be accommodated easily into most shoe types and potentially better tolerated when worn at night compared to currently available splints. Its design further allows it to be used comfortably during dynamic tasks such as walking and running as supported by initial anecdotal evidence in athletes. To date there has been no evaluation into the effectiveness of the DEFO in the general population with plantar fasciitis.

This study will look at the feasibility of conducting a randomised controlled trial into the use of a DEFO compared to an off-the-shelf orthoses as an adjunct to usual care.

DETAILED DESCRIPTION:
Plantar fasciitis is the most common foot and ankle pathology that affects the general population. It affects over 1 million people in the USA equating to ~0.2 million in the UK. It is characterized by severe pain felt on the plantar aspect of the heel around the plantar fascia origin which is significantly thicker than normal.

Usually conservative treatment comprises a referral to physiotherapy and provision of orthotics. Physiotherapy consists of teaching a home program of calf and plantar fascia stretches in addition to weight management and footwear advice.

Orthotic management includes the provision of off-the-shelf orthotics or customised orthotics. Some studies of customised orthoses demonstrate significant improvements in foot pain related function at 3 and 12 months in people with plantar fasciitis compared to a sham intervention. However, a systematic review of the randomised controlled trials found no evidence to support their use on short or long term foot pain, pain related function or disability.

Dynamic elastomeric fabric orthoses (DEFOs) have been successfully used in a variety of patient groups. The plantar fasciitis DEFOs is a custom-made close-fitting sock of elastomeric construction. It is worn next to the skin where the sock can exert an external torsional, compressive, and supportive effect, thus positively influencing the biomechanics of the heal.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Plantar heel pain for greater than 3 months

Exclusion Criteria:

* Calcaneal fracture
* Additional neurological or orthopaedic / rheumatological impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | Up to 12 weeks
  This is a patient reported questionnaire asking about the impact of the foot and ankle on 21 activities of daily living and 8-sport related activities. It has demonstrated validity for this client group (correlating with physical function subscales of the SF-36) and shows good test-retest reliability

SECONDARY OUTCOMES:
Visual Analogue scales | Up to 12 weeks
  Visual analogue / Numerical rating scales are commonly used to measure pain in clinical trials, having demonstrated good validity, reliability and responsiveness. Patients will indicate (a) their current heel pain and (b) their worst pain over the last 48 hrs using a numerical rating scale. 0 will indicate no pain at all and 10 will indicate their worst imaginable pain and numbers from 0-10 will be shown.
Ankle Range of Motion | Up to 12 weeks
  The extensibility of the ankle plantarflexors will be determined by measuring the angle of the tibia to the vertical using an inclinometer during a "lunge stretch".
Plantar Fascia thickness | Up to 12 weeks
  The thickness of the plantar fascia enthesis will be measured using ultrasound.
Quality of Life (QoL) | Up to 12 weeks
  This will be measured using both the Foot Health Status Questionnaire and the EQ-5D. The Foot Health Status Questionnaire measures foot health related quality of life and has demonstrated validity and reliability whilst the EQ-5D is recommended for health economic evaluations (and hence piloting of its use in this feasibility study is of value).

OTHER OUTCOMES:
Satisfaction | Up to 24 weeks
  A questionnaire, developed for the purposes of this study, will ascertain people's satisfaction with the DEFO/orthoses and their adherence over the previous week. This will be assessed 12 and 24 weeks (via post) after issuing the orthotic.
Participant characteristics | week 1
  The following patient characteristics and risk factors for the development of plantar fasciitis will be taken at baseline:
  * Age, gender
  * Duration of plantar fasciitis
  * Body mass index
  * Occupation and average hours standing per day
  * Physical activity (International Physical Activity Questionnaire
  * The number and type of hip / trunk exercises prescribed after the initial assessment by the treating therapist.
Recruitment and drop-out rates | Up to 24 weeks
  Data on recruitment and attrition rates will be entered into a database. Where possible, reasons for dropping out will be ascertained
  Percentage of completed measures at each time-point:
  The percentage of completed measures at each time-point for each participant will be entered onto a database
Feasibility | Up to 24 weeks
  At the end of the study participants and PHNT staff will complete a questionnaire on the feasibility of the study and provide suggestions that may aid the running of future trials
Effectiveness of blinding | Up to 12 weeks
  Following each measurement time point the assessor (RM) will be asked to indicate which group they think the participant was allocated to.
Cost | Up to 24 weeks
  Unit cost of each orthotic intervention (off-the-shelf orthotic Vs DEFO) will be gathered to help inform future economic evaluations. This will include an estimate of the time required to take the different measures required for fitting and ordering each orthosis.
Adherence | Up to 24 weeks
  A questionnaire, developed for the purposes of this study, will ascertain people's satisfaction with the DEFO/orthoses and their adherence to treatment over the previous week. This will be assessed 12 and 24 weeks (via post) after issuing the orthotic.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Marsden, PhD, Study Chair — Plumouth University; Richard McKee, B.Sc.(Hons), Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom